CLINICAL TRIAL: NCT00658281
Title: A Pilot Study of Setup Variation in the Supraclavicular Lymph Nodes Treatment in Breast Cancer Patients Using On-Board Imaging System With Linear Accelerator
Brief Title: Setup Variation in the Supraclavicular Lymph Nodes Treatment in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0132
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; On Board Imager Kilovoltage; Cone Beam Computed Tomography; Electronic Portal Imaging Device; Lymph Nodes; CBCT; OBI KV
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OBI KV System + CBCT Scanning: Breast cancer patient radiation treatment set up using OBI KV system and CBCT scanning or CT-on-rail system to verify standard EPID for positioning.
  Interventions: Procedure: CBCT Scan; Procedure: OBI KV Imaging

INTERVENTIONS:
Procedure: CBCT Scan — Cone Beam Computed Tomography (CBCT) scan performed once a week.
Procedure: OBI KV Imaging — On Board Imager kilovoltage (OBI KV) Imaging performed once a week.

SUMMARY:
The goal of this clinical research study is to use the On Board Imager kilovoltage (OBI KV) system and cone beam computed tomography (CBCT) scanning or CT-on-rail system to look at how well a routine device called an electronic portal imaging device (EPID) can set up a patient to receive radiation therapy on the lymph nodes in the neck.

DETAILED DESCRIPTION:
The Study Imaging Techniques for Radiation Treatment Planning:

The standard way to set up a patient to receive radiation therapy on the lymph nodes in the neck is by using an EPID, which uses high-energy X-rays to make images to see if the patient's body positioning for radiation therapy is correct or not. It is important for the doctors to see the position of the patient's lower neck so that radiation can be delivered to the right place.

The position of the patient's body during radiation therapy is typically checked once a week using an EPID or a similar device. While the patient is lying on the treatment table, the EPID system takes the necessary images. In this study, along with using an EPID, researchers will use the OBI KV system and CBCT scanning, in order to look at how well the standard EPID is describing the patient's neck position.

OBI KV imaging is designed to make images using low-energy X-rays, and the images are considered reasonably clear and easy for the doctors to read. CBCT scanning uses low-energy X-rays that let the doctors see the lymph nodes in the lower neck. Unlike regular CT scanning, CBCT scanning does not require "contrast" material to be used.

Since all 3 of the pieces of equipment (the EPID, OBI KV, and CBCT systems) are built into the same treatment machine, you will not need to move for the extra pieces of equipment that are being used in this study. You will lay very still, as usual, and the images will all be taken in a row.

Screening Tests:

The study doctor will review your medical chart to decide if you are eligible to take part in this study. If you are found to be eligible and you agree to take part, you will then begin the normal radiation treatment planning process. You will sign a separate consent form that will describe the radiation therapy and EPID procedures in more detail, as well as their risks.

During the treatment period when you are receiving radiation treatments once a day for 5 weeks, you will have CBCT scanning and OBI KV imaging performed once a week.

Before you receive radiation treatment, while you are lying on the treatment table, the EPID will be used. After that, the OBI KV and CBCT devices will rotate around you to take the images for this study. During the radiation therapy treatment, the EPID, OBI KV, and CBCT scans will be performed once a week, on the same day if possible. Sometimes the EPID and OBI KV scans will be performed during the same treatment, while the CBCT scan may be performed during another treatment that same week. It should take about 30 minutes to finish taking both the OBI KV and CBCT images.

The results of the CBCT scanning and OBI KV imaging will not, in any way, be used to plan your radiation therapy.

Length of Study Participation:

After your 5-week radiation treatment period, your participation in this study will be over.

This is an investigational study. The EPID is commercially available and FDA approved for use in setting up a patient to receive radiation therapy. OBI KV imaging and CBCT scanning are also commercially available and FDA approved for use in this purpose, but they are not typically used. What is experimental in this study is using additional procedures (OBI KV imaging and CBCT scanning) to check how reliably the EPID can set up a patient to receive radiation therapy on the lymph nodes in the neck.

Up to 30 evaluable patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed carcinoma of the breast.
2. American Joint Committee on Cancer (AJCC) Stage I-III, or locally recurrent breast cancer
3. Planned for radiation treatment of the supraclavicular and axillary apex nodal beds using a SCV field
4. Age greater than or equal to 18 years, since classic breast cancer is a disease of adults
5. Able to understand the current trial and give informed consent

Exclusion Criteria:

1. Has bilateral breast cancer requiring radiation to both breasts due to anatomic constraints on planning CT
2. inflammatory carcinoma due to altered treatment schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
System Failure (defined as 2 or more disagreements between the EPID and either OBI systems or CT-on-rail from among the 5 evaluations for a particular patient) | CBCT scanning and OBI R or CT-on-rial system, 5 evaluations per patient, during 5-week radiation treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Wang, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org